CLINICAL TRIAL: NCT04721847
Title: Effects of Pain Neuroscience Education in Diabetic Neuropathy
Brief Title: Pain Neuroscience Education in Diabetic Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/00752 Rameeza Warraich
Record Dates: First submitted 2021-01-19; First posted 2021-01-25 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Pain, Neuropathic; Diabetic Nephropathy
Keywords: Pain; Neuropathy; Diabetes
MeSH Terms: conditions — Neuralgia; Diabetic Nephropathies; Pain; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain Neuroscience Education (Experimental): Pain Neuroscience Education (PNE) sessions. Additionally, treated with Transcutaneous Electrical Nerve Stimulation (TENS), Stretching and Strengthening exercises similar as in control group
  Interventions: Other: Pain Neuroscience Education
- Conventional Physical therapy (Active Comparator): Control group will be treated by TENS, stretching and strengthening exercises.
  Interventions: Other: Conventional Physical therapy

INTERVENTIONS:
Other: Pain Neuroscience Education — In first part educational content will be designed to be given in group of patients in six sessions by PNE booklet. The six sessions are 1.5 hours long (9 hours) and will be given at a frequency of 1 session per week. Final session will be given to solve doubts, and to provide additional information to the educational program. Book for additional material will be delivered to participants.
  Arms: Pain Neuroscience Education
Other: Conventional Physical therapy — Control group will be treated by Conventional Physical therapy like TENS, stretching and strengthening exercises. Intervention will be initiated with warm up period (joint mobility exercises) for the duration of 5 mins and ended up with cool down period (relaxing exercises i.e. deep breathing) for the duration of 5 mins.
  Arms: Conventional Physical therapy

SUMMARY:
To determine the effects of Pain Neuroscience Education in Diabetic Neuropathy

DETAILED DESCRIPTION:
Pain neuroscience education (PNE) has shown to have immediate effects on various clinical signs and symptoms associated with central sensitization. Using a model of (innocuous, noxious and allodynia) PNE can be used in combination with exercise therapy, especially treating patients in which the nervous system has become increasingly hypervigilant. Teaching patients about the neuroscience of pain and lead to healthier and more positive attitudes and beliefs regarding chronic pain. Pain in diabetic neuropathy restrict the activity participation and compromise their quality of life. PNE will be helpful in such patients so decreasing pain can improve their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* History of diabetic ≥ 5 years
* HbA1C higher and equal to 6.5 %
* Self-completed Leeds Assessment of Neuropathic Symptoms and Signs pain scale (S-LANSS) ≥ 12
* Mini Mental State Examination (MMSE) score ≥ 24

Exclusion Criteria:

* Known neurological disorder
* Foot ulcers/candidate of amputation
* Hearing impaired

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2020-08-13 (Actual); Primary Completion 2021-07-28 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Numeric pain rating scale (NPRS) | 6 weeks
  The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable"). High test-retest reliability has been observed in both literate and illiterate patients with rheumatoid arthritis (r = 0.96 and 0.95, respectively) before and after medical consultation.
Self-completed Leeds Assessment of Neuropathic Symptoms and Signs pain scale (S-LANSS) | 6 weeks
  Total score is 24. If score < 12, neuropathic mechanisms are unlikely to be contributing to the patient's pain. If score ≥ 12, neuropathic mechanisms are likely to be contributing to the patient's pain. The S-LANSS has Cronbach α of .76 when completed unaided rising to α=.81 in neuropathic pain so this is reliable tool.

SECONDARY OUTCOMES:
Diabetic peripheral neuropathic pain impact measure | 6 weeks
  18 item DPNI is a reliable and valid Patient rating outcome measure disease impacts and treatment for DNP. Internal consistency ranged from 0.91 to 0.96 and test - retest from 0.84 to 0.91. All prespecified hypothesis for convergent and discriminant validity were met.

CONTACTS AND LOCATIONS:
Overall Officials: Mirza Obaid Baig, MSPT(NMR), Principal Investigator — Riphah International University
Locations (1):
- Allied Hospital, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No